CLINICAL TRIAL: NCT02283502
Title: For Research Purpose the Clinical Test of the Magnetic Resonance Imaging Guided Focused Ultrasound Ablation System on Uterine Fibroids
Brief Title: Clinical Test of the MRgHIFU System on Uterine Fibroids
Acronym: MRgHIFU
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chin-Jung Wang (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor-Investigator, Chin-Jung Wang, Associate Professor, MD, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHRI-CTC-067
Record Dates: First submitted 2014-10-28; First posted 2014-11-05 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-10

CONDITIONS: Uterine Fibroids
Keywords: Uterine fibroid; magnetic resonance imaging; ultrasound; non-invasive therapy
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention: MRgHIFU, Surgery (Experimental): Magnetic resonance-guided high-intensity focused ultrasound (MRgHIFU) system for the noninvasive treatment of uterine fibroids
  Interventions: Device: MRgHIFU system

INTERVENTIONS:
Device: MRgHIFU system — Magnetic resonance-guided high-intensity focused ultrasound (MRgHIFU) system for the noninvasive treatment of uterine fibroids

SUMMARY:
The objectives of this program are to verify the safety and effectiveness of the MRgHIFU system developed by the division of Medical Engineering of National Health Research Institutes (NHRI)

DETAILED DESCRIPTION:
Between 25 % - 50 % of women of childbearing age have uterine fibroids. Also, 25% of women with fibroids suffer from the metrorrhagia, menorrhagia, dysmenorrheal or pelvic compression so that they don't have a good quality of life. The worse case is the fertility of patients with fibroids is hindered. The current clinical treatment is medication or surgery. Medication can only suppress the symptom temporarily when the hysterectomy method of removing part or all of uterus can cure the patient completely. However, the hysterectomy is an invasive operation and the women with fibroids who plan to have a baby don't accept this kind of treatment.

Magnetic resonance-guided high-intensity focused ultrasound (MRgHIFU) system for the noninvasive treatment of uterine fibroids has been developed and was approved by the US Food and Drug Administration (FDA) in 2004. The ultrasound waves emitted by the ultrasonic probe propagate through the skin, fat, muscle, soft tissues and converge on fibroids at focus. High energy/intensity at focus causes the thermal necrosis of the fibroid tissue in several seconds. The whole process of HIFU ablation of fibroids is monitored and guided by MR thermometery. The advantage of MR-HIFU modality includes no incision, outpatient treatment and few side effects.

The objectives of this program are to verify the safety and effectiveness of the MRgHIFU system developed by the division of Medical Engineering of National Health Research Institutes (NHRI), to achieve the clinical trial at the Chang-Gung Memorial Hospitals of Linkou and to commercialize the self-developed MRgHIFU system. The mission is to conduct the first-stage clinical test for 10 women with symptomatic uterine fibroids and to make two sets of HIFU system. Meanwhile, the impact of quality of life and satisfaction with treatment of the patients diagnosed with symptomatic uterine fibroids will be analyzed.

ELIGIBILITY:
Inclusion criteria:

1. Already sign in the Informed Consent Form。
2. The woman who want to operate the Hysteromyomectomy, and the volume of the fibromyoma is between 5-10 cm, will be included。
3. Woman age between 35~45 years, and do not want to be pregnant
4. Abdominal circumference≦95 ㎝.
5. No pregnant.
6. MRI compatible.

Exclusion criteria:

1. Pregnant or Breast-feeding.
2. MRI uncompatible.
3. Woman who has scar in Abdomen.
4. Immunodeficiency or cancer.
5. Use the clinical medicine before 3 month age.
6. The woman who will not follow the project. -

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Check Adverse Event or Serious Adverse Event | six month
  follow up

SECONDARY OUTCOMES:
Using MRI to confirm the volume of the fibromyoma. | Screen, after treatment 1Month, 3Month, 6Month
  follow up difference of fibromyoma that before and after treatment
Using quality of life questionnaire to compare quality of life that before and after treatment | Screen, after treatment 1Month, 3Month, 6Month
  follow up

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Jung Wang, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Clinical Trial Center, Taoyuan District, Taiwan, Taiwan